CLINICAL TRIAL: NCT07267663
Title: Vein Wrapping in Peripheral Nerve Injury Repair Below The Elbow .
Brief Title: Vein Wrapping in Peripheral Nerve Injury Repair Below The Elbow
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Abd Elmoniem Mohamed, residant doctor at Assiut university hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vein Wrap in peripheral Nerve
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Nerve Injury Repair
Keywords: Vein Wrapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Active Comparator): patients will undergo standard epineural nerve repair with autologous vein wrapping, and outcomes will be assessed at follow-up intervals.
  Interventions: Procedure: nerve repair; Procedure: vien Wrapping

INTERVENTIONS:
Procedure: nerve repair — The nerve ends are repaired using a standard epineural microsuture technique (usually 8-0 or 9-0 nylon).
  Tension-free coaptation is ensured.
Procedure: vien Wrapping — The vein is wrapped loosely around the nerve repair site without any tension. The edges are sutured with a few fine 8-0 or 9-0 nylon stitches.

SUMMARY:
Peripheral nerve injuries are common after trauma and may cause pain, sensory loss, motor deficit, and long-term disability. Scar formation and perineural adhesion at the repair site interfere with axonal regeneration, impair gliding of the nerve within surrounding tissues, and are main contributors to painful neuroma formation and persistent functional deficits.

After peripheral nerve injury or incomplete regeneration, disorganized axonal sprouting and connective tissue proliferation at the proximal nerve end can result in a traumatic neuroma. This structure is characterized by tangled axons, Schwann cells, and fibrous tissue, leading to pain, hypersensitivity, and impaired function. Neuromas often develop when regenerating axons cannot reconnect with their distal targets, typically due to excessive scar formation or tension at the repair site.Scar tissue not only obstructs regenerating axons but also mechanically tethers the nerve, resulting in traction neuritis and painful hypersensitivity.

Autologous vein wrapping in which a segment of the patient's own vein is placed around the repaired nerve has been shown to reduce perineural scarring and neuroma formation by acting as both a mechanical barrier and a biological conduit. The vein sheath isolates the nerve from surrounding fibrotic tissue, while its inner endothelial surface supports axonal guidance and nutrient diffusion. Experimental studies have demonstrated improved axonal regeneration, reduced collagen deposition, and better functional recovery when vein wrapping is used compared to simple neurorrhaphy.

Clinical studies have also reported favorable outcomes with vein wrapping, particularly in preventing recurrent or painful neurom. It is a simple, cost-effective, and autologous technique that avoids immune reaction or foreign body response. Patients treated with vein wrapping often show reduced neuropathic pain and improved sensory recovery.

Clinically, Tinel's sign (Hoffmann-Tinel test) is widely used as a simple bedside test to detect regenerating axons advancing along a nerve or to localize symptomatic neuromas. A progressive distal-to-proximal Tinel's sign often indicates advancing regeneration, whereas a static or painful Tinel's sign at the repair or nerve ends may indicate neuroma-in-continuity or symptomatic end neuroma. Because it is easy to perform and commonly recorded in clinical follow-up, Tinel's sign is an appropriate secondary outcome to assess the presence of symptomatic neuroma or nerve regeneration after vein-wrapped repairs.

Therefore, this study aims to systematically evaluate the effect of autologous vein wrapping on neuroma formation, functional recovery, and associated clinical signs, such as Tinel's sign, in patients with traumatic peripheral nerve injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years with traumatic peripheral nerve injury requiring surgical repair.
* Nerve injury distal to the elbow.
* Time from injury to surgical repair less than 6 months .

Exclusion Criteria:

* Injury proximal to the elbow.
* Children below 18.
* History of multiple comorbidities (e.g., diabetes+another chronic illness)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of neuroma formation | 12 months postoperatively
  assessed by high-resolution ultrasonography

SECONDARY OUTCOMES:
Patient satisfaction and functional scores (DASH). | 12 months
  Patient satisfaction and functional scores (DASH).